CLINICAL TRIAL: NCT03646318
Title: Ketanserin Effects on Peripheral Temperature and Lactate (KoPTaL)
Brief Title: Ketanserin Effects on Peripheral Temperature and Lactate
Acronym: KoPTaL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, PHJ van der Voort, Prof. dr. P. H. J. van der Voort, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WO 17.123 oost
Record Dates: First submitted 2018-04-11; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Ketanserin

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial (blinded)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo medication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketanserin (Experimental): Ketanserin is a serotonin type 2-receptor blocker (5-HT2). In normal endothelium, the 5-HT1 effects (vasodilation) are the most prominent [Dabire 1990]. In endothelium that is damaged, which is the case in sepsis, the 5HT2 effects (vasoconstriction) surpass the 5-HT1 effects. Blocking the 5-HT2 receptor with ketanserin can attenuate this pathological vasoconstriction. In addition, ketanserin has favourable α1-adrenergic blocking properties in the endothelium (vasodilation) that may further reverse the pathological vasoconstriction. In these ways ketanserin can reduce vasoconstriction and can improve the microcirculation.
  Interventions: Drug: Ketanserin
- Placebo (Placebo Comparator): The placebo is a standard glucose 5% solution.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketanserin — The dose of 0.75 ug/kg/min is a dose that has been used frequently in critically ill patients. The concentration of the study drug infusion will be 40 mg/40 ml glucose 5%. The maximum dose however will be 4.5 mg per hour for patients with a weight more than 100 kg. The pre-filled 50 ml syringes will be filled with 40 ml of a solution containing 40 mg ketanserin or 0 mg ketanserin in glucose 5%.
  The minimum number of ketanserin vials (2 ml with 5 mg/ml) that are needed is 240 (40 mg = 4 vials per patient). Duration of intervention: 8 hours
  Arms: Ketanserin
Other: Placebo — Glucose 5% solution
  Arms: Placebo

SUMMARY:
A high blood lactate and a high peripheral to central temperature difference (deltaT) are associated with a higher mortality in critically ill patients. Both measures are signs of a reduced microcirculatory bloodflow or vasoconstriction and are associated with shock. It is unknown which medication can best be used to improve deltaT and lactate clearance.

Ketanserin is being used in the intensive care setting for decades to optimize circulatory parameters. Ketanserin is a serotonin type 2-receptor blocker (5-HT2). Blocking the 5-HT2 receptor with ketanserin can attenuate pathological vasoconstriction. In these ways ketanserin can reduce vasoconstriction and can improve the microcirculation. As a consequence, the enhanced blood flow in the skin will increase the peripheral temperature and decrease deltaT. At the same time an increased flow in the microcirculation may lead to a reduction in lactate production.

Objective:

To determine the effects of a continuous ketanserin infusion on peripheral temperature and lactate clearance in critically ill patients with either a high lactate or a high deltaT.

DETAILED DESCRIPTION:
Rationale:

A high blood lactate and a high peripheral to central temperature difference (deltaT) are associated with a higher mortality in critically ill patients. Both measures are signs of a reduced microcirculatory bloodflow or vasoconstriction and are associated with shock. On the other hand, it has not been shown yet that interventions leading to improvement of this temperature gap reduces mortality or improves any other outcome measurement. Moreover, it is unknown which medication can best be used to improve deltaT and lactate clearance.

Ketanserin is being used in the intensive care setting for decades to optimize circulatory parameters. Ketanserin is a serotonin type 2-receptor blocker (5-HT2). Blocking the 5-HT2 receptor with ketanserin can attenuate pathological vasoconstriction. In these ways ketanserin can reduce vasoconstriction and can improve the microcirculation. As a consequence, the enhanced blood flow in the skin will increase the peripheral temperature and decrease deltaT. At the same time an increased flow in the microcirculation may lead to a reduction in lactate production.

Objective:

To determine the effects of a continuous ketanserin infusion on peripheral temperature and lactate clearance in critically ill patients with either a high lactate or a high deltaT.

Study design:

A multicentre double blind randomized controlled trial.

Study population:

All adult intensive care patients above 17 years old with a deltaT of >6°C with informed consent given by the patient or legal representative.

Intervention (if applicable):

The intervention is a continuous pump driven Ketanserin infusion of 0.75 ug/kg/min for eight hours.

The control group will receive the same volume of glucose 5%.

Main study parameters/endpoints:

Change in DeltaT (measured per hour) Change in lactate (measured per 2 hours)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The risks of ketanserin infusion are limited but can be a QTc prolongation and a slight decrease in blood pressure. The study needs an arterial blood sample on inclusion, and after 2, 4, 6 and 8 hours of 1.5 ml each. In addition, a 6 ml blood sample at T=4 and T=8 hours.

ELIGIBILITY:
Inclusion Criteria:

* DeltaTemperature greater that 6.0 °C.
* Age 18 years or older
* Admitted to the ICU for any reason
* Signed informed consent from the patient or legal representative

Exclusion Criteria:

* Pregnancy
* No possibility to obtain informed consent
* QTc above 550 msec,
* Arrhythmias, including bradycardia defined as a heart rate below 50/min; 2nd and 3rd degree AV block; ventricular tachycardia
* Blood Potassium level < 3.5 mmol/l
* Blood Magnesium level <0.5 mmol/l
* Allergy for ketanserin
* DeltaT less than 6°C.
* Patients undergoing therapeutic hypothermia
* Patients admitted after cardiac arrest
* Patients admitted after cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Delta Temperature | 8 hours (after start of the study medication)
  Delta Temperature is calculated from the difference between central (rectal) and peripheral (forefoot) temperature

SECONDARY OUTCOMES:
Lactate clearance | 8 hours (after start of the study medication
  Lactate clearance is defined as :(Lactate (admission) - Lactate (8 hours))*100 / Lactate (admission) (Lactate (admission) - Lactate (8 hours))*100 / Lactate (admission) A lactate clearance of 10% or more is regarded as clinical relevant
hospital length of stay | 6 months after start of study medication
  Length of stay hospital
mortality | 6 months after start of study medication
  mortality at hospital discharge
ICU length of stay | 6 months after start of study medication
  length of stay in the ICU
ICU mortality | 6 months after start of study medication
  mortality at ICU discharge

IPD SHARING:
Plan to Share IPD: No